CLINICAL TRIAL: NCT02662621
Title: Pilot Study With the Aim to Quantify a Stress Protein in the Blood and in the Urine for Early Diagnosis of Malgnant Solid Tumors
Brief Title: Pilot Study With the Aim to Quantify a Stress Protein in the Blood and in the Urine for the Monitoring and Early Diagnosis of Malignant Solid Tumors
Acronym: EXODIAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: INSERM U866 Faculté de Médecine et Pharmacie (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A01638-39
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cancer
Keywords: personalized care; early diagnosis; ovarian cancer; breast cancer; lung cancer; Early Detection; Cancer [E01.390.500]
MeSH Terms: conditions — Neoplasms; Disease; Ovarian Neoplasms; Breast Neoplasms; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ill patient (Other): Patient with a cancer disease
  Interventions: Other: blood samples; Other: Urine samples
- Healthy volunter (Other): Subject without any cancer pathology
  Interventions: Other: blood samples; Other: Urine samples

INTERVENTIONS:
Other: blood samples
Other: Urine samples

SUMMARY:
Recent studies shows that extracellular vesicles (named "exosomes") released by cancer cells exhibit at their membrane the stress protein HSP70, contrary to exosomes released by normal cells. These exosomes ("HSP70-exosomes") have a very important role in intercellular communication and have specific biological functions that can promote tumor progression. They are found in the different biological fluids such as blood and urine.

We have developed a protocol able to isolate exosomes in blood and urine. We also demonstrated that only exosomes derived from cancer cell have HSP70 at their membrane. Those results strongly suggest that we can only identify exosomes with HSP70 at the membrane in patients with cancer.

Detection of HSP70-exosomes in the diagnosis of patients is a promising pathway of research. Because a cancer cell can releases a large amount of exosomes (several billion) and since its appearance, our approach will allow to earlier detect cancer with respect to the use of imaging and circulating tumor cells (CTCs), which remains a rare event (about one CTC of 1 billion cells).

The aim of this study is to demonstrate that HSP70-exosomes could be used for early diagnosis of patients with malignant solid tumor. In order to demonstrate this, the objective of the study is to study blood and urine samples from 60 subjects with a malignant tumor and 20 healthy subjects (witness).

ELIGIBILITY:
Inclusion criteria for patients

* Women newly diagnosed with either:
* Infiltrating non-metastatic breast cancer (positive or negative HER2 status or hormone therapy)
* Breast cancer with a first metastasis evolution (positive or negative HER2 status or hormone therapy).
* Ovarian cancer stage III and IV,
* Men and women who are newly diagnosed non-small cell lung cancer metastatic,
* Age ≥18 years
* Affiliation to a social security system,
* Signed Informed consent.

Exclusion Criteria for patients:

* Patient with another synchronous tumor,
* Men with breast cancer,
* Positive HIV and / or HBV and / or HCV serology
* Patients unable to undergo a medical monitoring for geographical, social or psychological condition,
* Pregnant or nursing women,
* People enjoying a major protection system (including trusteeship and guardianship).

Inclusion criteria for healthy volonter

* Men or women aged 50-70 years (mean age of onset of various cancers in the study)
* Affiliation to a social security system,
* Signed Informed consent.

Exclusion criteria for healthy volonter

* history of cancer,
* Positive HIV and / or HBV and / or HCV serology
* Pregnant or nursing women,
* People enjoying a major protection system (including trusteeship and guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
concentration of HSP70 exosomes in the blood and urine | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ISAMBERT, MD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- CGFL, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chanteloup G, Cordonnier M, Isambert N, Bertaut A, Marcion G, Garrido C, Gobbo J. Membrane-bound exosomal HSP70 as a biomarker for detection and monitoring of malignant solid tumours: a pilot study. Pilot Feasibility Stud. 2020 Mar 3;6:35. doi: 10.1186/s40814-020-00577-2. eCollection 2020. PMID 32161659